CLINICAL TRIAL: NCT03302546
Title: Incremental Hemodialysis as a Starting Way of Renal Replacement Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 034/17
Record Dates: First submitted 2017-07-03; First posted 2017-10-05 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incremental Hemodialysis (Active Comparator): Subjects on this arm will be treated with 2 hemodialysis sessions of at least 4 hour per week.
  Interventions: Procedure: Incremental hemodialysis
- Conventional hemodialysis (Active Comparator): Subjects on this arms will be treated with 3 hemodialysis sessions of at least 3.5 hour per week.
  Interventions: Procedure: Conventional hemodialysis

INTERVENTIONS:
Procedure: Incremental hemodialysis — Patients randomized to this arm of treatment will be treated during at least 4 hours of hemodialysis twice per week
  Arms: Incremental Hemodialysis
Procedure: Conventional hemodialysis — Patients randomized to this arm of treatment will be treated during at least 3.5 hours of hemodialysis three times per week
  Arms: Conventional hemodialysis

SUMMARY:
The Hemodialysis Unit of the Hospital Ramon y Cajal is a pioneer in the implementation of a program of incremental hemodialysis, starting with two sessions a week in patients with residual renal function.

The main objective is to compare whether the initiation of hemodialysis with two sessions a week over conventional pattern of initiation of three sessions a week better preserves residual renal function.

DETAILED DESCRIPTION:
The primary specific objective is to assess the loss of renal function defined as 24 hours diuresis less than 100 ml at 12 months of starting treatment. Secondary objectives are: erythropoietin dose, concentration of beta 2-microglobulin, p-cresol, fenol, the state of hydration and nutrition, adverse effects, hospital admissions, mortality and quality of life, comparing both arms of treatment.

DESIGN: Multicenter randomized clinical trial. Randomization will be performed by an external agent that guarantees an homogeneous balance between both arms. The randomization sequence will not be available for the investigators responsible of the patients.

Inclusion criteria: Patients starting hemodialysis that maintain residual diuresis and urea clearance greater than or equal to 2.5 ml / min with a minimum follow-up of one year.

Exclusion criteria: Anuric patients, patients with acute renal failure and patients who start hemodialysis after having going through a renal transplant.

The variables that will be analyzed are 24h diuresis, urea clearance, creatinin clearance, haemoglobin, leukocytes, platelets, creatinin, urea, Na, K, albumin, prealbumin, Ca, P, PTH, PCR, ferritin, B2microglobulin, BNP, KT/V, Erythropoietin dose, state of hydratation and life quality.

Sample size should be of 42 patients on each arm of treatment to obtain a 95% confidence (α=0,05) and a 80% of statistical power (β=0,20).

The normality of the data will be analyzed with Kolmogorov-Smirnov test which will allow to use parametric tests (T-student) or non-parametric tests (U-Mann-Whitney). Association of categoric variables of both arms will be analyzed with Chi2 test, or using Fisher statistic.

Loss of renal function will be analyzed up to 12 months and time studies will be performed through non-parametric test (Kaplan-Meier), obtaining the estimated probability of loss of renal function in both arms and comparing survival functions through "Log-Rank" statistic.

The demonstration of efficacy and safety through a clinical trial would spread this clinical practice in the nephrology community and therefore in our national health system.

ELIGIBILITY:
Inclusion Criteria:

* Subjects starting renal replacement therapy from January 2017 to June 2018.
* Subjects who consent to sign the Informed Consent Form.
* Subject who maintain residual diuresis and urea clearance equal or superior to 2,5 ml/min.

Exclusion Criteria:

* Anuric patients.
* Patients with acute renal failure.
* Patients who revoke the Informed Consent Form.
* Patients who start hemodialysis after having going through a renal transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Asses the loss of residual renal function in patients who started chronic hemodialysis | Measurements of multiple variables to measure renal function each two months during one year period
  Assess the loss of renal function evolution in patients starting hemodialysis therapy 2 days per week, versus patients with hemodialysis 3 days per week.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain

REFERENCES:
- [Derived] Fernandez Lucas M, Ruiz-Roso G, Merino JL, Sanchez R, Bouarich H, Herrero JA, Muriel A, Zamora J, Collado A. Initiating renal replacement therapy through incremental haemodialysis: Protocol for a randomized multicentre clinical trial. Trials. 2020 Feb 19;21(1):206. doi: 10.1186/s13063-020-4058-0. PMID 32075665